CLINICAL TRIAL: NCT06446830
Title: The Analgesic Efficacy of Vitamin B Complex with Paracetamol and Non-steroidal Antiinflammatory Medication in Critically Ill Obstetrics After Caesarian Section; a Prospective Randomized , Placebo-controlled and Double-blinded Study
Brief Title: The Analgesic Efficacy of Vitamin B Complex in Critically Ill Obstetrics After Caesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R370/2023
Record Dates: First submitted 2024-06-02; First posted 2024-06-06 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Analgesia; Post Operative Pain; Cesarean Section
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: two parallel-group, randomized, double-blinded
Who Masked: Participant, Outcomes Assessor
Masking Description: the candidate will be masked, and Assessments regarding the primary outcome will be conducted by an assessor blind to treatment allocation. The assessor will go through a profound assessment training program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin B (Experimental): oral vitamin B complex tablets preoperative and continue post-operative for 2 days One tablet oral once daily for 1- 2 days according to the length of stay; the tablet is a vitamin (B1, B6, B9, and B12).
  Oral daily vitamin B concentration; Tablet is composed of ; B1= 250mg, B6= 150 mg, B12= 0,250 mg, B9= 0.5mgm, B2 15 mg standard analgesic ladder will be implemented in the form of; Paracetamol 1gram (2 tablets) / 8hr for 48 hours, Ketorolac 30 mg / 12 hour for 48 hours. Any pain will be treated appropriately with nalbuphine till the patient is comforted, and the total dose will be documented.
  the routine ladder of paracetamol and ketorolac will be modified according to organ functions and the presence of any contraindication for usage
  Interventions: Drug: multimodal analgesia and vitamin B
- standard (Active Comparator): patients will receive a preoperative; Oral placebo tablet (once/day) Post-operative and continue post-operative for 2 days; One placebo capsule oral once daily for 2 days. standard analgesic ladder will be implemented in the form of; Paracetamol 1 gram (2 tablets) / 8hr for 48 hours. Ketorolac / 12 hours for 48 hours. Any pain will be treated appropriately with nalbuphine till the patient is comforted, and the total dose will be documented.
  the routine ladder of paracetamol and ketorolac will be modified according to organ functions and the presence of any contraindication for usage
  Interventions: Drug: standard multimodal analgesia

INTERVENTIONS:
Drug: multimodal analgesia and vitamin B — B1, B6 , B9 , B12 in addition to the routine paracetamol and NSAID
  Other Names: neuroton tablets
  Arms: vitamin B
Drug: standard multimodal analgesia — Routine Paracetamol and NSAID
  Arms: standard

SUMMARY:
We aim to investigate the value of vitamin B (B1, B6, B9, B12) on post-cesarean section analgesia in addition to the standard opioid-sparing multimodal regimen to achieve more robust analgesia with minimal side effects.

DETAILED DESCRIPTION:
Optimum analgesia is an essential component in enhanced recovery after elective and emergency Caesarean section. Opioid-based analgesia negatively affects maternal functional recovery. Unlike other types of surgeries, the performance and the quality of postoperative recovery in caesarean section affects two individuals: the patient and their infant, hence it is recommended to use Opioid-sparing medications post-caesarean section.

Multimodal analgesia is recommended for post-caesarean section pain control. The main properties of its components are to promote return of (i) Mobility (ii) Oral intake (iii) Normal bowel function (iv) Micturition: Trial without urinary catheter (v) Activities of daily living, with Few adverse effects: inactive metabolites (no nausea, vomiting, sedation, pruritus, constipation or respiratory depression), Readily available after discharge home, Little risk of dependency (especially long-term opioids), Minimal risk of hyperalgesia or chronic pain and cost-efficient with minimally invasive technique and no side-effects on the neonate.

The morbidity of critically ill obstetrics can increase due to inadequate control of pain and also due to the consumption of opioid analgesia due to associated respiratory depression, sedation, and nausea. Multimodal analgesia is strongly recommended.

An immune-histochemistry study found that B vitamins potentiate acute morphine antinociception. In other studies, the value of vitamin B complex on postoperative analgesia was discussed and investigated in different combinations Another study reported the value of folic acid in decreasing gastric hypersensitivity in maternal stress in rats. Other studies explained the benefit of folic acid in analgesia through modulating gut microbiota, reducing inflammation, modulating purinergic signaling, and promoting nerve repair (6)This is the first study to investigate the effect of vitamin B9 (folic acid ) and other vitamin B (B1, B6, B12) beside the standard opioid sparing analgesics on post-caesarean section pain in critically ill obstetrics.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill -obstetric patients who will be delivered by cesarean section under neuraxial anesthesia.

Exclusion Criteria:

1. Patient's Refusal to participate
2. Known allergy to one or more of the given components.
3. Disturbed conscious level.
4. Prolonged or complicated surgery; defined by operative time of more than 90 min.
5. Severe liver dysfunction or failure
6. Severe renal dysfunction or failure.
7. Severe thrombocytopenia; platelets less than 50

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-25 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The total consumption of rescue analgesics in the first and second 24 hours after delivery | in the first 24 hours and in the second 24 hours (if stay is extended )
  the difference in mean of the total amount consumed of paracetamol, ketorolac and nalbuphine
Pain score assessed by numerical pain scale after 24 hours from delivery. | 24 hours postoperative
  By using a s scale from 0-10 where zero is no pain and 10 is the worst pain, the scale willbe used 24 hours postoperative . results will be compared between both groups

SECONDARY OUTCOMES:
quality of recovery on discharge from ICU | on discharge from ICU ( or within 48 hours post operative ) which is shorter
  using The Obstetric Quality of Recovery-10A questionnaire where less than 70 will be considered poor recovery , and the higher the score will be linked to better recovery
occurrence of any side effects | during ICU stay and no more than 48 hours post-caesarean section
  occurrences of any side effects as allergy

CONTACTS AND LOCATIONS:
Overall Officials: wessam selima, MD, Principal Investigator — assistant professor (lecturer)- Ain shams university
Locations (1):
- Ain shams university, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dautzenberg B, Truffot-Pernot C, Hazebroucq J, Legris S, Guerin C, Begelman C, Guermonprez G, Fievet MH, Chastang C, Grosset J. A randomized comparison of two clarithromycin doses for treatment of Mycobacterium avium complex infections. Infection. 1997 Jan-Feb;25(1):16-21. doi: 10.1007/BF02113501. PMID 9039532
- [Background] Deng XT, Han Y, Liu WT, Song XJ. B Vitamins Potentiate Acute Morphine Antinociception and Attenuate the Development of Tolerance to Chronic Morphine in Mice. Pain Med. 2017 Oct 1;18(10):1961-1974. doi: 10.1093/pm/pnw358. PMID 28379583
- [Background] Moskowitz DB. Marketplace. How the stock market fall hits health care firms. Faulkner Grays Med Health. 1997 Nov 3;51(43):suppl 2 p.. No abstract available. PMID 10173708
- [Background] Wong TC, Lai MM. Avian reticuloendotheliosis virus contains a new class of oncogene of turkey origin. Virology. 1981 May;111(1):289-93. doi: 10.1016/0042-6822(81)90674-7. No abstract available. PMID 6263007